CLINICAL TRIAL: NCT01457170
Title: Investigating the Acute Pulmonary Vascular Haemodynamic Effects of Apelin in Pulmonary Hypertension
Brief Title: Effects of Apelin on the Lung Circulation in Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: NHS Lothian (Other Government); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11/CARD/04
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Arterial Hypertension; Heart Failure
Keywords: Pulmonary Hypertension; Heart Failure; Apelin; Haemodynamics; pulmonary vascular resistance; cardiac output
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Failure; Hypertension, Pulmonary | interventions — Apelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apelin/Saline (Experimental): Apelin infusion then crossover to Saline infusion
  Interventions: Drug: Apelin; Drug: Saline (Placebo)
- Saline/Apelin (Experimental): Saline infusion then crossover to Apelin infusion
  Interventions: Drug: Saline (Placebo); Drug: Apelin

INTERVENTIONS:
Drug: Apelin — During right heart catheterisation, Apelin will be infused at 30, 100 and 300 nanomol/min for 5 minutes. Apelin will then be infused at 300 nanomol/min for a further 15 minutes while the subject exercises using a supine ergometer.
  Arms: Apelin/Saline
Drug: Saline (Placebo) — During right heart catheterisation, saline will be infused for 15 minutes while the subject rest and for a further 15 minutes while the subject exercises using a supine ergometer.
  Arms: Apelin/Saline
Drug: Saline (Placebo) — During right heart catheterisation, saline will be infused for 15 minutes while the subject rest and for a further 15 minutes while the subject exercises using a supine ergometer.
  Arms: Saline/Apelin
Drug: Apelin — During right heart catheterisation, Apelin will be infused at 30, 100 and 300 nanomol/min for 5 minutes. Apelin will then be infused at 300 nanomol/min for a further 15 minutes while the subject exercises using a supine ergometer.
  Arms: Saline/Apelin

SUMMARY:
The purpose of this study is to determine the effects of Apelin on the lung circulation. The investigators hypothesise that Apelin will relax the lung blood vessels and improve the pumping ability of the heart.

DETAILED DESCRIPTION:
Apelin is an endogenous peptide with physiological actions in the cardiovascular system and is abundantly expressed in the pulmonary vasculature. Pre-clinical models and preliminary clinical data indicate that Apelin deficiency may mediate or contribute to the pathogenesis of pulmonary hypertension and heart failure. Apelin causes peripheral vasodilatation and increased cardiac contractility. The investigators will determine the effects of Apelin on the pulmonary circulation in 3 groups; healthy control, people with pulmonary arterial hypertension and people with pulmonary hypertension due to heart failure. Each subject will receive both Apelin infusion and saline placebo infusion in a crossover design. The infusions will be given in a random order which the subject and the investigator will be blinded to. The investigators hypothesise that Apelin will have more marked pulmonary haemodynamic effects than that observed in the systemic circulation. Moreover, the investigators propose that Apelin will have a marked vasodilatory effect on the human pulmonary vasculature and reduce pulmonary vascular resistance in patients with pulmonary arterial hypertension or pulmonary hypertension due to left heart disease.

ELIGIBILITY:
PULMONARY ARTERIAL HYPERTENSION

Inclusion Criteria:

* Pulmonary Arterial Hypertension which is Idiopathic, Heritable, associated with connective tissue disease or associated with drugs/toxins
* mean pulmonary artery pressure >/= 25mmHg
* pulmonary capillary wedge pressure < 15 mmHg
* normal/reduced cardiac output
* stable
* WHO functional class II - IV

Exclusion Criteria:

* significant left ventricular dysfunction
* chronic lung disease (FEV1 < 60% or abnormal CT)
* chronic thromboembolic pulmonary hypertension

HEART FAILURE

Inclusion Criteria:

* stable on treatment for 3 months prior to study
* NYHA grade II - IV
* ejection fraction <35%, left ventricular end-diastolic diameter > 5.5 cm and/or shortening fraction < 20%
* Tricuspid regurgitant velocity >/= 3.0 m/s

HEALTHY VOLUNTEERS

Inclusion Criteria:

* mean pulmonary artery pressure < 25 mmHg
* tricuspid regurgitant velocity < 2.5 m/s

Exclusion Criteria:

* obstructive coronary artery disease

ALL SUBJECTS

Exclusion Criteria:

* bleeding diathesis
* women of childbearing potential without pregnancy test
* systolic blood pressure > 190 mmHg or < 100 mmHg
* malignant arrhythmias
* renal or hepatic failure
* haemodynamically significant valvular heart disease
* severe or significant co-morbidity
* pacemaker
* already taking part in another trial
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance | 5,10,15 and 30 minutes after start of infusion
  We will measure the change in pulmonary vascular resistance after infusion of Apelin during right heart catheterisation

SECONDARY OUTCOMES:
Change in systemic vascular resistance | 5,10,15 and 30 minutes after start of infusion
  We will measure the change in systemic vascular resistance during infusion of Apelin
Change in Cardiac Output | 5,10,15 and 30 minutes after start of infusion
  We will measure the change in cardiac output after infusion of Apelin during right heart catheterisation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Peacock, BSc MPhil MD, Principal Investigator — National Health Service: Golden Jubilee National Hospital
Locations (3):
- United Kingdom (3):
  - Royal Infirmary Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Brash L, Barnes GD, Brewis MJ, Church AC, Gibbs SJ, Howard LSGE, Jayasekera G, Johnson MK, McGlinchey N, Onorato J, Simpson J, Stirrat C, Thomson S, Watson G, Wilkins MR, Xu C, Welsh DJ, Newby DE, Peacock AJ. Short-Term Hemodynamic Effects of Apelin in Patients With Pulmonary Arterial Hypertension. JACC Basic Transl Sci. 2018 Mar 28;3(2):176-186. doi: 10.1016/j.jacbts.2018.01.013. eCollection 2018 Apr. PMID 29876530